CLINICAL TRIAL: NCT00041665
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Trial of Recombinant Human Keratinocyte Growth Factor for Reduction of Mucositis in Patients With Hematologic Malignancies Undergoing Total Body Irradiation and High-dose Chemotherapy With Autologous PBPC Transplantation
Brief Title: Recombinant Human Keratinocyte Growth Factor to Reduce Oral Mucositis in Hematologic Malignancy Patients Undergoing Peripheral Blood Stem Cell Transplantation After Radiation and High-dose Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20000162; NLM Identifier NCT00020813; UCLA-0012064; MSKCC-01065; FHCRC-161200; NCT00020813 (obsolete NCT alias)
Record Dates: First submitted 2002-07-11; First posted 2002-07-15 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Stomatitis
MeSH Terms: conditions — Stomatitis | interventions — Fibroblast Growth Factor 7

INTERVENTIONS:
Drug: Recombinant Human Keratinocyte Growth Factor

SUMMARY:
Radiotherapy and high dose chemotherapy with bone marrow transplantation or peripheral blood stem cell transplantation is frequently used as treatment for patients with cancers of the bone marrow or lymph nodes such as Hodgkin's disease, non-Hodgkin's lymphoma, leukemia or multiple myeloma. A common side effect of the radiotherapy and high dose chemotherapy is mucositis (inflammation of the inside of the mouth and throat resulting in pain and difficulty swallowing). Mucositis is often very severe such that patients receive intravenous nutrition and pain medication in the hospital.

In this study, an investigational recombinant human growth factor called Keratinocyte Growth Factor (rHuKGF) is being evaluated to determine its protective effect on the mucosal tissue and its ability to reduce the mouth and throat soreness.

ELIGIBILITY:
Inclusion Criteria: * Patients with: non-Hodgkin's lymphoma, Hodgkin's disease, acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic lymphocytic leukemia, or multiple myeloma * Eligible for fractionated total body irradiation (fTBI) plus high-dose chemotherapy followed by autologous PBPC support. * 18 years of age or older * Karnofsky performance status greater than or equal to 70% * Minimum of 1.5 Mio CD34+ cells/kg cryopreserved and to be transplanted * Informed consent for participation in the study Exclusion Criteria: * History of, or concurrent cancer other than NHL, Hodgkin's disease, AML, ALL, CML, CLL, multiple myeloma * Prior bone marrow or peripheral blood stem cell transplantation * Purged stem cell product * Currently active infection or oral mucositis * Congestive heart failure * Serum creatinine > 1.5x ULN * Direct bilirubin > 1.5x ULN * Transaminases > 3x ULN * Corrected DLCO < 50% of predicted * Subject is currently enrolled in, or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving other investigational agent(s). * Subject is pregnant (eg, positive human chorionic gonadotropin [HCG] test) or is breastfeeding. * Subject refuses to use adequate contraceptive precautions. * Known hypersensitivity to any of the products to be administered during dosing, including E coli-derived products. * Inability to give a truly informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Stiff PJ, Emmanouilides C, Bensinger WI, Gentile T, Blazar B, Shea TC, Lu J, Isitt J, Cesano A, Spielberger R. Palifermin reduces patient-reported mouth and throat soreness and improves patient functioning in the hematopoietic stem-cell transplantation setting. J Clin Oncol. 2006 Nov 20;24(33):5186-93. doi: 10.1200/JCO.2005.02.8340. Epub 2006 Jan 3. PMID 16391299
- [Result] Elting LS, Shih YC, Stiff PJ, Bensinger W, Cantor SB, Cooksley C, Spielberger R, Emmanoulides C. Economic impact of palifermin on the costs of hospitalization for autologous hematopoietic stem-cell transplant: analysis of phase 3 trial results. Biol Blood Marrow Transplant. 2007 Jul;13(7):806-13. doi: 10.1016/j.bbmt.2007.03.004. Epub 2007 Apr 23. PMID 17580258
- [Result] Stiff PJ, Erder H, Bensinger WI, Emmanouilides C, Gentile T, Isitt J, Lu ZJ, Spielberger R. Reliability and validity of a patient self-administered daily questionnaire to assess impact of oral mucositis (OM) on pain and daily functioning in patients undergoing autologous hematopoietic stem cell transplantation (HSCT). Bone Marrow Transplant. 2006 Feb;37(4):393-401. doi: 10.1038/sj.bmt.1705250. PMID 16415901
- [Result] Spielberger R, Stiff P, Bensinger W, Gentile T, Weisdorf D, Kewalramani T, Shea T, Yanovich S, Hansen K, Noga S, McCarty J, LeMaistre CF, Sung EC, Blazar BR, Elhardt D, Chen MG, Emmanouilides C. Palifermin for oral mucositis after intensive therapy for hematologic cancers. N Engl J Med. 2004 Dec 16;351(25):2590-8. doi: 10.1056/NEJMoa040125. PMID 15602019
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com